CLINICAL TRIAL: NCT04528264
Title: Ultrasound Guided Closed Reduction of Depressed Zygomatic Arch Fractures Compared to Conventional Blind Reduction: A Randomized Double Blind Clinical Trial
Brief Title: Ultrasound Guided Closed Reduction of Depressed Zygomatic Arch Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: College of Medical Sciences Teaching Hospital. Nepal (Other)
Responsible Party: Principal Investigator, Ashutosh Kumar Singh, Associate Professor, College of Medical Sciences Teaching Hospital. Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMSNepal
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Zygomatic Arch Fracture
Keywords: zygomatic arch fracture; Intraoperative Imaging; guided reduction

STUDY DESIGN:
Intervention Model Description: Randomized double blind
Who Masked: Participant, Outcomes Assessor
Masking Description: Sealed Envelope will be used to conceal allocation. Patients will be unaware of their group allocation. Outcome assessor will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided (Experimental): Intraoperative high frequency ultrasound used to guide the reduction of depressed zygomatic arch.
  Interventions: Device: Intraoperative ultrasound guided
- Conventional blind reduction technique (Other): Conventional blind reduction of zygomatic arch fracture will be conducted without any intraoperative imaging.
  Interventions: Other: Conventional blind reduction technique

INTERVENTIONS:
Device: Intraoperative ultrasound guided — Samsung Mysono U6 machine with LN 15 linear (https://www.samsunghealthcare.com/en/products/UltrasoundSystem/MySono%20U6/General%20Imaging/transducers) probe capable of Musculoskeletal imaging will be used for visualization and location of fracture after which elevation and reduction of fracture will be attempted. The ultrasound probe will be used as described by McCann. Radiographic continuity of periosteal shadow without any step will be taken as end point for reduction and the procedure will be terminated.
  Other Names: Intraoperative USG Imaging
  Arms: Ultrasound guided
Other: Conventional blind reduction technique — Conventional blind reduction technique
  Other Names: comparator
  Arms: Conventional blind reduction technique

SUMMARY:
Zygomatic arch fractures have always been treated with blind closed reduction and is the most commonly used method. Blind reduction of fractures might lead to inadequate reduction and associated complications of facial asymmetry and limitations in mouth opening which may require reoperation for correction. Various methods like portable CT scan, C arm fluoroscopy, endoscopy and ultrasound have been proposed and used to visualize the reduction for better outcome. Out of these, ultrasound is inexpensive, easily available, easy to use, non-ionizing and has greatest potential to be used as standard for visual reduction of zygomatic arch fractures. There are studies where ultrasound has been compared to blind method and other modalities but level I evidence and recommended protocol for its intraoperative use has been lacking.

DETAILED DESCRIPTION:
Isolated and depressed zygomatic arch fractures have an incidence of about 5 to 14% of lateral mid face fractures. Depressed zygomatic arch fractures have been managed by blind closed reduction historically based upon tactile sense of surgeon and auditory click assumed as the conclusive evidence of reduction. The minimal fracture exposure for zygomatic arch fractures either solitary or combined with zygomaticomaxillary complex fractures results in inadequate visibility of the fractures and inadequate or inappropriate reduction of fractures. These fractures can be visualized by surgical exposure with coronal approach but is limited by complications and extensive training required. Other options are intraoperative imaging with portable CT scan but they are cumbersome, require radiologists for positioning and are not available in all operative units as well as expensive. Endoscopic visualization and reduction are another option for intraoperative control of these fractures but endoscopes are expensive, not available in all operative units and require experience and training to use appropriately. Various studies and our own experience show that unacceptable number of depressed zygomatic arch fractures remain incompletely reduced with blind reduction method. The resulting deficit might be as small as a depressed lateral face, inadequate sagittal projection of cheek to inadequate mouth opening. Portable ultrasound machines are readily available in almost all anesthesia units and operating rooms. These ultrasound units can be utilized to reduce the zygomatic arch satisfactorily with real time image guidance and it has advantage of being radiation free and inexpensive compared to fluoroscopy based portable C arm units. A small pilot in our own unit has shown remarkable difference between reduction achieved under ultrasonography guidance vs closed reduction based on tactility. This method should be explored and perfected to bring in common use among Oral & Maxillofacial surgeons so that blind assumption of fracture reduction is replaced by a more scientific confirmation of fracture reduction.

ELIGIBILITY:
Inclusion Criteria:

* 6 years and above
* fractured and depressed zygomatic arch requiring surgical reduction

Exclusion Criteria:

* pregnant patients
* not willing for participation
* below 6 years age

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Post operative radiographic evidence of adequate reduction | 24 hours
  The radiographic evaluation will be performed blinded by one of the clinician oral and maxillofacial surgeons who will not be involved in any of the operations. The adequacy of reduction will be evaluated in a DICOM viewing software on axial scans to assess contour of the arch and step if any at the fracture site.
  1. Good reduction : Absence of any step and straight contour of zygomatic arch symmetric to contralateral uninjured arch
  2. Average reduction: Absence of any step but poor contour of zygomatic arch and asymmetric to contralateral uninjured arch
  3. Poor reduction: Presence of both a cortical step and asymmetric arch compared to contralateral uninjured arch
Facial profile symmetry | one week to four weeks
  Clinical assessment will be performed blinded by a clinician oral and maxillofacial surgeon who will not be involved in any of the operations on first postoperative day, first follow up visit after one week of operation and 4 weeks of operation. Facial symmetry and projection will be assessed clinically by the clinician and graded as good, adequate and poor. A patient oriented clinical outcome is considered good practice and clinically relevant in modern evidence based medicine so patient response will be recorded as binary (yes/no) response regarding their view on facial symmetry.
Number of reoperations | 24 hours
  Revision surgery required after failed reduction assessed and confirmed radiographically on CT scan and clinical assessment as well as patient reported measure of facial symmetry and adequate mouth opening.
Mouth opening | at 24 hours postoperatively
  Interincisal opening measured between the incisal tips of central incisor teeth and recorded in millimeter using a vernier caliper.

SECONDARY OUTCOMES:
Operative time | Intraoperative
  Additional time required to reduce with intervention.
Number of attempts or reduction | Intraoperative
  Additional attempts required with imaging guidance.
Cost of intervention | Intraoperative
  Additional cost required with imaging guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh K Singh, MDS, Principal Investigator — College of Medical Sciences, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Fully sharable link will be provided after study completion with deidentified data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after completion and publication
Access Criteria: Decided by PI
URL: https://www.researchgate.net/project/USG-guided-closed-reduction-of-depressed-zygomatic-arch-fractures

REFERENCES:
- See also: Project page on Researchgate — https://www.researchgate.net/project/USG-guided-closed-reduction-of-depressed-zygomatic-arch-fractures